CLINICAL TRIAL: NCT00902993
Title: A Phase I, Randomised, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD1446 in Male and Non-fertile Female, Young and Elderly Healthy Volunteers, After Oral Multiple Ascending Doses
Brief Title: Study to Investigate Safety, Tolerability and Pharmacokinetics With Single and Multiple Ascending Doses of AZD1446
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D1950C00002; EudraCT No. 2008-008389-10
Record Dates: First submitted 2009-05-12; First posted 2009-05-15 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
Keywords: MAD; NNR; to investigate safety and tolerability in a multiple ascending dose study in Healthy subjects; AZD1446
MeSH Terms: interventions — 3-(5-chloro-2-furoyl)-3,7-diazabicyclo(3.3.0)octane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Part A single and multiple dose and part B fractionated dose
  Interventions: Drug: AZD1446
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1446 — Solution, oral single and multiple dose
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
This study is designed to evaluate the safety, tolerability and PK of AZD1446 in Subjects when given as multiple dose administration for either 7 Days (Day 1 single dose, Day 2-6 multiple doses) in Part A and optionally at fractionated doses for 1 Day in Part B.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-fertile female, young or elderly Subjects, aged ≥18 to ≤50 or ≥65 to ≤80
* Body mass index (BMI) between 19 and 30 kg/m2
* Clinically normal findings on physical examination

Exclusion Criteria:

* History of any clinically significant disease or disorder
* History of severe allergy/hypersensitivity reactions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-04; Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Part A: to assess the safety and tolerability of AZD1446 following multiple ascending doses of an orally administered solution of AZD1446 in male and non-fertile female, young and elderly Healthy Volunteers, | during the whole study period, ca 50 days
Part B: to assess the safety and tolerability of AZD1446 following administration of an oral solution of AZD1446 as fractionated doses during one day in male and non-fertile female, young and elderly Healthy Volunteers. | during the whole study period, ca 43 days

SECONDARY OUTCOMES:
Part A: To determine the single and multiple dose PK of AZD1446 in male and non-fertile female Healthy Volunteers. | PK sampling taken at defined timepoints during residential period, 10 days for Part A and 4 days for Part B
Part B: To mimic an extended release dosing regimen and determine the fractionated dosing PK of AZD1446 in male and non-fertile Healthy Volunteers. | PK sampling taken at defined timepoints during residential period, 10 days for Part A and 4 days for Part B

CONTACTS AND LOCATIONS:
Overall Officials: Björn Paulsson, MD, PhD, Study Director — AstraZeneca; Marianne Hartford, MD PhD, Principal Investigator — AstraZeneca Clinical Pharmacology Unit (CPU) Sahlgrenska University Hospital GöteborgSE-413 45 GöteborgSweden; Ingemar Bylesjo, MD PhD, Principal Investigator — AstraZeneca Clinical Pharmacology Unit (CPU) C2:84Karolinska University Hospital HuddingeSE-141 86 StockholmSweden
Locations (2):
- Sweden (2):
  - Research Site, Gothenburg
  - Research Site, Stockholm